CLINICAL TRIAL: NCT01585454
Title: Healthy Lifestyle in Pregnancy
Status: Withdrawn | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999912108; 12-DK-N108
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2016-01-20

CONDITIONS: Hperglycemia; Diabetes Mellitus; Weight Gain
Keywords: Pregnancy; Diabetes Mellitus; Weight Gain; Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Women can gain too much weight or develop diabetes during pregnancy. If the mother is overweight or has diabetes during pregnancy, her baby may also be at risk of being overweight or developing diabetes. A woman s chance of getting diabetes increases if her parents or family members are overweight or have diabetes. Poor diet and exercise habits can also lead to weight gain and diabetes. Researchers want to study how best to improve the health of pregnant women and their children. They will do so by providing healthy lifestyle counseling for women receiving prenatal care at the Phoenix Indian Medical Center.

Objectives:

- To study the effectiveness of healthy lifestyle counseling for overweight and/or diabetic pregnant women.

Eligibility:

* Women at least 18 years of age who will receive pregnancy care at the Phoenix Indian Medical Center.
* Participants must be overweight or obese. They may or may not have diabetes.

Design:

* Participants will receive standard prenatal care from the midwives, doctors, and dietitians at the Phoenix Indian Medical Center.
* Participants will work with National Institutes of Health staff for about 2 hours every week. These sessions may include phone calls, home visits, or group meetings.
* Participants will have a total of nine measurement visits. The first visit will be at or before 16 weeks of pregnancy. The next three visits will be within a week of the first visit. Another four visits will take place between 23 and 28 weeks of pregnancy.
* Participants will have different tests through their pregnancy. They will wear heart monitors and wrist monitors to measure heart rate and movement. They will provide information on their eating habits, physical activity, and mood and feelings during pregnancy. Blood samples will be collected to measure blood glucose (sugar) levels.
* Participants will receive counseling on healthy eating and physical activity habits. They will be encouraged to invite friends or family members to learn more about healthy lifestyle choices.
* The study will end with the final visit about 6 to 8 weeks after giving birth. A final blood sample will be collected. Participants will be asked questions about mood and feelings.

DETAILED DESCRIPTION:
American Indians are at high risk for developing type 2 diabetes mellitus (T2DM) and its complications. Major factors responsible for this finding include obesity and intrauterine exposure to diabetes; the latter increases the risk of diabetes in the offspring particularly during childhood and adolescence. This study is designed to evaluate the feasibility of conducting an intensive lifestyle intervention (ILI) in adult (age greater than or equal to 18 years) pregnant women of any race or ethnicity who are eligible for prenatal care at Phoenix Indian Medical Center (PIMC). Most of these women or their fetuses will be of American Indian heritage. Interventions will be provided to overweight and obese pregnant women who may have diabetes, develop gestational diabetes (GDM), or be at high risk of developing diabetes. We will evaluate our ability to maintain engagement and motivate adoption of a healthy diet and increased physical activity. The lifestyle intervention will be patterned after the Diabetes Prevention Program (DPP) that prevented or delayed the onset of diabetes in non pregnant adults; the interventions will be modified to be appropriate in pregnancy. A major modification will be to encourage managed weight gain instead of weight loss. For women who have or develop diabetes, interventions will include coaching to optimize glycemic control. In this protocol, we will seek to identify strategies that can successfully accomplish these goals. Results from this study will permit us to formulate appropriate intervention strategies for a large randomized clinical study to evaluate the impact of an intensive lifestyle intervention on pregnant women and their offspring.

The project will be conducted in collaboration between the nurse midwifery and obstetrics services at Phoenix Indian Medical Center (PIMC) and the National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK). Important feasibility measures include evaluating our ability to enroll and retain pregnant women in a lifestyle intervention program and collect serial measures of gestational weight and glucose, objective measures of physical activity, and nutritional questionnaires.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. At least 18 years of age.
  2. Receive prenatal care at the nurse midwifery/obstetrics service of PIMC and plan to continue receiving such care throughout the pregnancy.
  3. Are able to have an OGTT prior to 16 weeks gestation (if diabetes was not previously diagnosed). Hyperemesis can preclude some pregnant women from successfully completing the OGTT; these women will not be excluded if the fasting blood samples can be obtained. Pregnant women with previously diagnosed diabetes are eligible if measures of glycemia (FPG, HbA1c, glycated albumin) are completed prior to 16 weeks gestation.
  4. Estimated prenatal BMI >25 kg/m2.
  5. Able to commit the time required for the interventions and follow-up.
  6. Able and willing to provide informed consent.

EXCLUSION CRITERIA:

1. Contraindication to aerobic or resistance exercise (ACOG, 2002).
2. Twin or multiple gestation.
3. Severe anemia, uncontrolled asthma, uncontrolled hypertension, cardiac disease, or any condition that requires follow-up at specialty care clinics outside of PIMC (e.g., pregnancies at high risk for maternal or fetal demise).
4. Any condition that in the opinion of the investigators would interfere with consent, treatment, or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03-27; Study Completion 2016-01-20

PRIMARY OUTCOMES:
Gestational Weight Gain

SECONDARY OUTCOMES:
Gestational Diabetes
Complications of Pregnancy and Delivery

CONTACTS AND LOCATIONS:
Overall Officials: William C Knowler, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)

REFERENCES:
- [Background] Cedergren MI. Optimal gestational weight gain for body mass index categories. Obstet Gynecol. 2007 Oct;110(4):759-64. doi: 10.1097/01.AOG.0000279450.85198.b2. PMID 17906006
- [Background] Dabelea D, Hanson RL, Lindsay RS, Pettitt DJ, Imperatore G, Gabir MM, Roumain J, Bennett PH, Knowler WC. Intrauterine exposure to diabetes conveys risks for type 2 diabetes and obesity: a study of discordant sibships. Diabetes. 2000 Dec;49(12):2208-11. doi: 10.2337/diabetes.49.12.2208. PMID 11118027
- [Background] International Association of Diabetes and Pregnancy Study Groups Consensus Panel; Metzger BE, Gabbe SG, Persson B, Buchanan TA, Catalano PA, Damm P, Dyer AR, Leiva Ad, Hod M, Kitzmiler JL, Lowe LP, McIntyre HD, Oats JJ, Omori Y, Schmidt MI. International association of diabetes and pregnancy study groups recommendations on the diagnosis and classification of hyperglycemia in pregnancy. Diabetes Care. 2010 Mar;33(3):676-82. doi: 10.2337/dc09-1848. No abstract available. PMID 20190296